CLINICAL TRIAL: NCT00397488
Title: Phase II Study of Sunitinib in Metastatic Transitional Cell Carcinoma of the Urothelium
Brief Title: Sunitinib in Treating Patients With Progressive Metastatic Transitional Cell Cancer of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-081; MSKCC-06081
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; anterior urethral cancer; posterior urethral cancer; recurrent urethral cancer; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Sunitinib

ARMS (1):
- Sunitinib (Experimental): This is a phase II trial of Sunitinib in patients with metastatic urothelial carcinoma. Sunitinib will be administered at a dose of 50 mg orally once daily for four consecutive weeks followed by a two-week rest period for the initial population. A second cohort of patients will be enrolled, who will receive 37.5 mg of sunitinib orally, on a continuous dosing schedule. Intra-patient dose reduction may be required depending on the type and severity of individual toxicity encountered. Re-staging imaging studies will be performed after every cycle of treatment during the first 4 cycles and subsequently after every other cycle. Patients may continue on study as long as they are tolerating therapy and in the absence of disease progression.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with progressive metastatic transitional cell cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with progressive metastatic transitional cell carcinoma of the urothelium treated with sunitinib malate.
* Determine the safety of this regimen in these patients.

Secondary

* Determine the time to disease progression in patients treated with this regimen.

  * To determine time to tumor progression (TTP) for sunitinib malate on a continuous dosing schedule for treatment of metastatic urothelial carcinoma.
  * To estimate sunitinib and SU012662 trough plasma concentration (Ctrough) data for the continuous daily schedule and to determine potential association with efficacy and safety.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the urothelium, including 1 of the following sites:

  * Bladder
  * Urethra
  * Ureter
  * Renal pelvis
* Progressive metastatic disease

  * Progressive disease defined as new or progressive lesions on cross-sectional imaging
  * Progressed despite prior treatment with cytotoxic chemotherapy
* Measurable disease
* Previously treated disease, as defined by the following:

  * Received treatment with 1-4 cytotoxic agents
  * Prior therapy must have included ≥ 1 of the following:

    * Cisplatin
    * Carboplatin
    * Paclitaxel
    * Docetaxel
    * Gemcitabine hydrochloride
  * Prior cytotoxic agents in the perioperative or metastatic setting allowed and may have been administered sequentially (e.g., first-line treatment followed by second-line treatment at time of progression) or all as part of a single regimen
* No symptomatic CNS metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin ≤ 1.5 mg/dL (unless Gilbert's disease is present)
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver function abnormalities are due to underlying malignancy)
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* None of the following within the past 6 months:

  * Myocardial infarction
  * Severe or unstable angina
  * Coronary or peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* No ongoing cardiac dysrhythmias ≥ grade 2
* No prolonged QTc interval on baseline ECG
* No uncontrolled hypertension, defined as blood pressure > 150/100 mm Hg despite optimal medical therapy
* No preexisting thyroid abnormality (i.e., thyroid function tests that cannot be maintained in the normal range with medication)
* No known HIV- or AIDS-related illness or other active infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy or chemotherapy
* At least 4 weeks since prior major surgery
* No other concurrent investigational drugs
* No concurrent participation in another clinical trial (supportive care trials or non-treatment trials [e.g., quality of life] allowed)
* No concurrent therapeutic doses of warfarin (low-dose warfarin ≤ 2 mg once daily for thromboembolic prophylaxis allowed)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean F. Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Sunitinib in patients with metastatic urothelial carcinoma.
Period: Overall Study
Arm/Group | Sunitinib
Started | 78
Completed | 71
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Response rate as measured by RECIST criteria. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). In general, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 71
participants
  Partial Response (PR) | 3
  Stable Disease (SD) | 29
  Progression of Disease (POD) | 39

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 34/78
Other Adverse Events (participants affected / at risk) | 67/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=78)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Death not associated with CTCAE term- Death NOS (General disorders) | 4 (4)
Death not associated with CTCAE term-Disease progression (General disorders) | 2 (2)
Dehydration (General disorders) | 2 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Extremity-lower (gait/walking) (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Fistula, GI- Small bowel (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Bladder infection (Renal and urinary disorders) | 2 (2)
Sepsis (General disorders) | 1 (1)
Pneumonia (General disorders) | 1 (1)
Infection (Infections and infestations) | 4 (4)
Memory impairment (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Pain - Back (General disorders) | 3 (3)
Pain - Bone (General disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 2 (2)
Pain - Head/headache (General disorders) | 2 (2)
Pain - Pelvis (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=78)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 8 (8)
ALT, SGPT (Blood and lymphatic system disorders) | 5 (5)
Anorexia (General disorders) | 4 (4)
AST, SGOT (Blood and lymphatic system disorders) | 6 (6)
Creatinine (Metabolism and nutrition disorders) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 28 (28)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 18 (18)
Heartburn/dyspepsia (Gastrointestinal disorders) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 28 (28)
Hemorrhage, Urinary NOS (Renal and urinary disorders) | 5 (5)
Hypertension (Cardiac disorders) | 6 (6)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 29 (29)
Lymphopenia (Blood and lymphatic system disorders) | 19 (19)
Nausea (Gastrointestinal disorders) | 7 (7)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 20 (20)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 7 (7)
Platelets (Blood and lymphatic system disorders) | 20 (20)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (5)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 5 (5)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 13 (13)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 5 (5)
Weight loss (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes